CLINICAL TRIAL: NCT01743209
Title: A Retrospective Non-interventional Descriptive Epidemiology Study for Patients With Paraphilia Sex Offenders Receiving Androgen Antagonists Treatment
Brief Title: Descriptive Epidemiology Study for Patients With Paraphilia Sex Offenders and Receiving Androgen Antagonists
Acronym: EPIPARA
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2012/057/HP
Record Dates: First submitted 2012-12-04; First posted 2012-12-06 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Paraphilia
Keywords: androgen antagonists
MeSH Terms: conditions — Paraphilic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The main objective of the study is to describe the french population of individuals with paraphilia who have committed a sexual offence in whom androgen antagonists was prescribed. The secondary objectives are the description of social demographic profiles, the personal and family histories,psychiatric co-morbidities, the side effects of androgen antagonists treatment. This study, the first of its kind in France, may allow to better understand the social demographic and clinical profile of sexual offenders with paraphilias treated with androgen antagonists.

To be included, the subject must have committed a sexual offense and must present a diagnosis of paraphilia with an indication of treatment with androgen antagonists. Paraphilia is defined by the Diagnostic and Statistical Manual as a sexual behavior disorder characterized by "sexually arousing fantasies, needs or recurrent and intense sexual behaviors generally involving (1) of non-human objects, (2) the suffering or humiliation of oneself or partner, (3) children or other persons without their consent, occurring during a period of at least six months "(Criterion A). This disorder is responsible for sexual behavior which is "clinically significant disturbances in social, occupational or other important areas of functioning" (Criterion B).

The inclusion of approximately 200 subjects is expected in this study. The inclusion period will last for 12 months.

Data will be codified and only a few investigators will have access to these data. The statistical analyse will use the usual descriptive parameters: mean, standard deviation, median, interquartile range and range for quantitative variables, frequencies and cumulative frequencies (if applicable) for qualitative variables.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of paraphilia based on DSM-IV-TR
* antecedent of sexual offence

Exclusion Criteria:

* no diagnostic of paraphilia

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients sex offenders with paraphilia and treatment with androgen antagonists
Sampling Method: Non-Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2012-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
current deviant sexual activity assessed with the frequency of deviant sexual activity per month | first visit (day 1)
  The primary outcome measure concerns the patient current deviant sexual activity. These data are reported routinely by the patient during his medical consultation and consigned in the medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Florence THIBAUT, MD/PhD, Principal Investigator — University Hospital, Rouen; Heloise Delavenne, MD, Study Chair — University Hospital, Rouen; Sandrine LAMY, MD, Study Chair — University Hospital, Rouen
Locations (1):
- University Hospital of Rouen, Rouen, France